CLINICAL TRIAL: NCT04318964
Title: An Open, Single Arm and Early Clinical Study of TAEST16001 in the Treatment of Solid Tumor Mainly Containing Soft Tissue Sarcoma With Positive Expression of Tumor Antigen NY-ESO-1 (HLA-A * 02:01)
Brief Title: TAEST16001 in the Treatment of Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Xiangxue Precision Medical Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xing Zhang, Vice director of department of medical sarcoma and melanoma,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-senU-TAEST16001
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAEST16001 cells treat tumor antigen NY-ESO-1 (Experimental): The dose escalation was carried out according to the principle of "3 + 3" increase. Four dose levels (calculated by the number of tcr-t positive cells) were set up: the dose level was 1: 5 × 108 ± 30%; the dose level was 2: 2 × 109 ± 30%; the dose level was 3: 5 × 109 ± 30%; the dose level was 4: 1.2 × 1010 ± 30%. Three patients in the first group, if there is no DLT, they will be enrolled in the next higher dose group; if one of the three patients in a certain dose group has DLT, three patients in the group will be supplemented with the same dose and method. If DLT occurred in 1 or more of the 3 cases, the dose increase was stopped. The former dose was defined as MTD; if DLT did not occur in 3 cases, the dose increased to the next group. Dose escalation is not allowed for the same patient.
  Interventions: Biological: TAEST16001 cells

INTERVENTIONS:
Biological: TAEST16001 cells — The patients in the dose increasing part and the expanding part received the intravenous reinfusion of TAEST16001 cells on the 5th day (i.e. the interval was 4 days) after the lymphocyte elimination chemotherapy: If the dose level of reinfusion was 1 and 2, the planned total amount of TAEST16001cells (calculated by TCR-T positive cells) was given a single reinfusion on the 1st day of the study. If the dose level of reinfusion was 3 and 4,then the total amount of TAEST16001cells (calculated by TCR-T positive cells) was planned to be reinjected in 60% and 40% proportion on the first and second day of the study.
  After the first reinfusion of TAEST16001 cells, the patients will be given a small dose of IL-2 subcutaneously (study day 1 to day 14), 500000 U / time. The first injection will be carried out within 30 minutes after the cell reinfusion, twice a day (interval 10-12 hours), for 14 days.

SUMMARY:
This study is an open, single arm, dose increasing early clinical study, which is divided into two parts: "3 + 3" designed dose escalation study and extended group study. The purpose of this study is to evaluate the safety, tolerance, PK, PD characteristics, and preliminary efficacy of TAEST16001 immunotherapy in the treatment of patients with solid tumor maily containing soft tissue sarcoma whose tumor antigen NY-ESO-1 expression is positive (HLA-A * 02:01).

DETAILED DESCRIPTION:
Immunotherapy is one of the most promising and effective methods to cure tumor besides operation, chemotherapy and radiotherapy. T cell therapy, which belongs to immunotherapy, mainly includes CAR-T (Chimeric Antigen Receptor, CAR) and TCR-T (T cell Receptor-T). The existing CAR-T treatment can only kill blood tumor cells, the effect on solid tumor treatment was not well. Therefore, people need a better method than CAR-T, which can kill tumor cell internal antigen and has better curative effect on solid tumor treatment, and has less side effect. This is the TCR-T cell treatment developed by the applicant now.

In view of the cross reaction between tumor antigen and normal cell antigen, which is easy to cause adverse reactions, this mainly focuses on a kind of antigen that is not expressed in normal cells, but expressed in testis, and is defined as cancer testis antigen. The applicant preferred NY-ESO-1 antigen, which was first found in esophageal cancer, then 10-50% in melanoma, non-small cell lung cancer (NSCLC), liver cancer, breast cancer, prostate cancer, bladder cancer, thyroid cancer and ovarian cancer, 60% in multiple myeloma, 70-80% in synovial cell sarcoma and 22.5% in osteosarcoma.

In 2015, the University of Pennsylvania, the University of Maryland and Adaptimmune in the United Kingdom reported the breakthrough progress of TCR-T cells in the world-class Journal of natural medicine. This clinical trial showed that high affinity anti-NYESO-1 and LAGE-1 specific TCR-T were effective in 16 (80%) of 20 patients with multiple myeloma, with an average progression free survival of 19.1 months, and the side effects were mild, without serious side effects of CAR-T.

Another clinical trial of NY-ESO-1-specific TCR-T in the treatment of synovial cell sarcoma (synovial cell sarcoma) and melanoma by a team of Dr. Rosenberg from the National Cancer Research Institute of the United States showed that 61% of synovial cell sarcomas and 55% of melanoma had clinical effects. Due to the good clinical results of anti-NY-ESO-1-specific TCR-T of adaptimmune company in the treatment of synovial sarcoma, the US FDA approved this TCR-T cell treatment of synovial sarcoma to enter the breakthrough treatment

These clinical data indicate that TCR-T cell therapy can be applied to a variety of tumors, including soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent form (ICF) (genotype and tumor antigen screening and primary screening) should be signed before any research related operation;
2. Age ≥ 18 years and ≤ 70 years;
3. Advanced solid tumor with definite pathological diagnosis;
4. Unresectable advanced solid tumor that fails to undergo standard treatment (disease progression or recurrence or intolerable, such as chemotherapy, radiotherapy, targeted treatment, etc.) or lacks effective treatment:

1) Soft tissue sarcoma: a) Soft tissue sarcoma failed to be treated by chemotherapy containing doxorubicin and ifosfamide; 2) Primary liver cancer: a) Child Pugh liver function score A within 7 days before cell reinfusion; 3) Ovarian cancer: a) Platinum based chemotherapy (such as paclitaxel combined with carboplatin) failed. 4) Non small cell lung cancer (NSCLC): a) failure (disease progression or toxicity intolerance) or lack of effective treatment method of previous standard treatment (including platinum chemotherapy scheme or driven gene targeted treatment); 5) Breast cancer: a) patients who have received standard treatment failure or not applicable standard treatment.

5、At least 1 measurable lesion (according to recist1.1 standard） 6、Genotype and tumor antigen screening must meet the following two criteria: 1) HLA-A * 02:01 positive; 2) NY-ESO-1 positive: immunohistochemistry positive cells ≥ 20%; 7、ECOG score 0-1 and expected survival time > 3 months; 8. Color Doppler echocardiography indicates left ventricular ejection fraction ≥ 50%; 9. Laboratory test results should at least meet the following criteria:

* White blood cell count ≥ 3.0 × 109 / L
* Absolute neutrophil count (ANC) ≥ 1.5 × 109 / L (without the support of G-CSF and GM-CSF, at least 14 days before CLT);
* Absolute lymphocyte count (ALC) ≥ 0.7 × 109 / L;
* Platelet (PLT) ≥ 75 × 109 / L (no transfusion treatment 14 days before CLT);
* Hemoglobin ≥ 10g / dl (no transfusion treatment 14 days before CLT);
* Prothrombin time international INR ≤ 1.5 × ULN, unless anticoagulant therapy is used;
* APTT ≤ 1.5 × ULN, unless anticoagulant therapy is used;
* Serum creatinine ≤ 1.5mg/dl (or 132.6 μ mol / L)
* Creatinine clearance ≥ 60ml / min;
* AST / SGOT ≤ 2.5 × ULN; - ALT / SGPT ≤ 2.5 × ULN; - TBIL ）≤1.5×ULN； 10、Women of childbearing age who have not undergone sterilization before menopause must agree to use effective contraceptive measures within one year from the beginning of study treatment (chemotherapy for clearing lymph nodes) to the end of cell transfusion, and the serum pregnancy test is negative within 14 days before the first cell transfusion.

  11、Men who have not undergone sterilization must agree to use effective contraceptive measures from the beginning of the study treatment (chemotherapy) until one year after the last cell transfusion.

Exclusion Criteria:

1. The last dose of anti-tumor therapy (chemotherapy, endocrine therapy, targeted therapy, immunotherapy, tumor embolization or traditional Chinese medicine / Chinese herbal medicine with anti-tumor indications) was received within 4 weeks before cell reinfusion;
2. The live attenuated vaccine had been inoculated within 4 weeks before cell reinfusion;
3. The patients with bone metastasis in the whole body;
4. It is known that any component used in the treatment of this study will produce allergy Response;
5. Not recovered from previous operation or treatment-related adverse reactions to < 2-level CTCAEv5.0;
6. Patients with a history of meningeal or central nervous system metastasis, or patients with clear basic diseases of central nervous system and left significant symptoms within 6 months before cell transfusion;
7. Patients with poor drug control hypertension (systolic blood pressure > 160mmhg and / or diastolic blood pressure > 90mmHg) or with clinical significance Cardiovascular and cerebrovascular diseases, such as cerebrovascular accident (within 6 months prior to signing the master informed consent), myocardial infarction (within 6 months prior to signing the master informed consent), unstable angina pectoris, congestive heart failure with NYHA grade II or above, or serious arrhythmia that cannot be controlled by drugs or has potential impact on research and treatment Results of ECG showed clinically significant abnormality or average QTCF ≥ 450ms;
8. Combined with other serious organic or mental diseases;
9. Suffering from systemic active infection requiring treatment, including but not limited to active tuberculosis, known HIV positive patients or clinical active hepatitis A, B and C Patients with inflammation, including virus carriers, should be excluded;
10. Patients with autoimmune diseases: those with inflammatory bowel disease history and those with autoimmune disease history determined by the researchers as unsuitable for this study, such as systemic lupus erythematosus, vasculitis, and invasive lung disease, should be excluded (except vitiligo subjects);
11. Those with cell transfusion within 4 weeks before and during the study should be used (if there is a long-term plan) Use) systemic sterols, hydroxyurea, immunomodulators (e.g., interferon α or γ, GM-CSF, mTOR inhibitors, cyclosporin, thymosin, etc.);
12. History of organ transplantation, allogeneic stem cell transplantation, and renal replacement therapy;
13. Diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or liver failure that are not known to be controlled;
14. Alcohol and / or drug abusers;
15. Pregnant or lactating women;
16. Subjects with any coexisting medical conditions or diseases that may affect the development of this study determined by the investigator;
17. Subjects without legal capacity / limited capacity of behavior;
18. Patients who have received similar gene therapy products within 4 weeks before cell reinfusion and are not suitable for inclusion by evaluation;
19. Patients judged by the investigator are difficult to complete all visits or procedures required by the protocol (including the follow-up period), or insufficient compliance to participate in the study, or the patients considered unsuitable by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose (MTD） | Time Frame: From cell infusion up to 28 days
  MTD was defined as the previous lower dose of DLT in ≥ 2 / 6 patients.
Dose limited toxicity (DLT) | Time Frame: From cell infusion up to 28 days
  Adverse events associated with cell therapy are identified by the safety review board (SRC)

SECONDARY OUTCOMES:
Peripheral blood TAEST16001 cell peak (C Max) | From cell infusion up to 28 days
  The maximum concentration of TAEST16001 cells observed in peripheral blood. TAEST16001 cells were detected by flow cytometry and TCR-T DNA was detected by qPCR.
Peripheral blood TAEST16001 cell peak time (T Max) | From cell infusion up to 28 days
  The time required to observe maximum concentration of TAEST16001 cells in peripheral blood, TAEST16001 cells were detected by flow cytometry and TCR-T DNA was detected by qPCR.
Peripheral blood TAEST16001 cell AUC 0-28 | From cell infusion up to 28 days
  Area under the Concentration-time Curve from Zero up to a Definite Time Day 28
T cell subsets | From cell infusion up to 28 days
  5mL venous blood was collected and sent to the center laboratory for flow cytometry.
Peripheral blood antigen-specific CTL | From cell infusion up to 28 days
  5mL venous blood was collected and sent to the center laboratory for flow cytometry of cytotoxic T Cell.
Effector cell activity | Within 2 hours before leukocyte apheresis, 1 hour after the first cell infusion (study day 1), and on study days 7, 28, 60, 90, 180, 270.
  5mL venous blood was collected and sent to the center laboratory for enzyme-linked immunosorbent spot (ELISPOT) assays to evaluate the number of PBMC cells secreting cytokines, such as IFN-γ, IL-6, TNF-α, etc.
Objective response rate (ORR) | At baseline, on day 28, day 60, day 90, day 180, and day 270 after TAEST16001 cell infusion.
  The proportion of patients who achieved a confirmed partial response or complete response (RECIST 1.1 criteria).
Disease control rate (DCR) | At baseline, on day 28, day 60, day 90, day 180, and day 270 after TAEST16001 cell infusion.
  The proportion of patients who reached an objective response or stable disease (RECIST 1.1 criteria).
Progression free survival (PFS) | At baseline, on day 28, day 60, day 90, day 180, and day 270 after TAEST16001 cell infusion.
  The time interval from patient enrollment to disease progression (PD) (RECIST 1.1 criteria) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Zhang, professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Xing Zhang, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Pan Q, Weng D, Liu J, Han Z, Ou Y, Xu B, Peng R, Que Y, Wen X, Yang J, Zhong S, Zeng L, Chen A, Gong H, Lin Y, Chen J, Ma K, Lau JYN, Li Y, Fan Z, Zhang X. Phase 1 clinical trial to assess safety and efficacy of NY-ESO-1-specific TCR T cells in HLA-A *02:01 patients with advanced soft tissue sarcoma. Cell Rep Med. 2023 Aug 15;4(8):101133. doi: 10.1016/j.xcrm.2023.101133. PMID 37586317